CLINICAL TRIAL: NCT07043257
Title: The Effect of Escape Room-Based Bladder Catheterization Training on Nursing Students' Academic Achievement, Problem-Solving Skills, and Motivation: A Mixed-Methods Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Tugce Kabak Solak, TKSOLAK, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AGRSABFTKS002
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: NURSING EDUCATION; NURSING STUDENTS; ESCAPE ROOM; BLADDER CATHETERIZATION
Keywords: NURSING EDUCATION; BLADDER CATHETERIZATION; ESCAPE ROOM; MOTIVATION; PROBLEM-SOLVING SKILLS

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escape Room-Based Training (Experimental): Nursing students in this group will receive bladder catheterization training using an escape room-based educational method. The intervention includes problem-solving tasks, scenario-based puzzles, and gamified steps that reinforce clinical knowledge and psychomotor skills related to catheterization procedures.
  Interventions: Behavioral: Escape Room-Based Bladder Catheterization Training
- Traditional Training (Other): Nursing students in this group will receive traditional bladder catheterization training based on lecture-based theoretical instruction and standard simulation practice without gamified or interactive components.
  Interventions: Behavioral: Traditional Bladder Catheterization Training

INTERVENTIONS:
Behavioral: Escape Room-Based Bladder Catheterization Training — This intervention involves an escape room-based educational strategy designed to teach bladder catheterization to nursing students. The method includes interactive puzzles, clinical problem-solving tasks, and scenario-based simulations. The training promotes engagement, teamwork, and application of theoretical knowledge in a gamified learning environment.
  Arms: Escape Room-Based Training
Behavioral: Traditional Bladder Catheterization Training — This intervention includes standard bladder catheterization training based on traditional teaching methods. The students will receive theoretical instruction through lectures and demonstration-based simulation without interactive or gamified components.
  Arms: Traditional Training

SUMMARY:
This study aims to examine the effect of escape room-based training on nursing students' academic achievement, problem-solving skills, collaborative learning, and motivation levels in bladder catheterization education. A mixed-methods design will be used. Participants will be randomly assigned to either an experimental group receiving game-based escape room training or a control group receiving traditional instruction. Pre-test and post-test assessments will be conducted using validated measurement tools. The study also includes qualitative data to explore students' experiences and perceptions regarding the educational method used. This research seeks to contribute to innovative educational practices in nursing skills training.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students enrolled in a clinical skills course
* Voluntarily agree to participate
* No prior formal catheterization training

Exclusion Criteria:

* Students who miss training sessions
* Students with previous experience in escape room-based learning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-07-05 (Estimated)

PRIMARY OUTCOMES:
Academic Achievement | At Baseline, immediately after the intervention
  Academic achievement will be measured using a researcher-developed theoretical and practical knowledge test on bladder catheterization. The test includes multiple-choice and skill-based items aligned with clinical guidelines. Higher scores indicate greater knowledge and procedural competence.
Problem-Solving Ability | At Baseline, immediately after the intervention
  Problem-solving skills will be assessed using the Problem Solving Inventory (Heppner & Petersen). This validated scale measures students' perceptions of their problem-solving ability. Higher scores indicate lower perceived problem-solving ability (reverse scoring will be considered in interpretation).
Motivation Level | At Baseline, immediately after the intervention
  Students' motivation will be measured using the Motivation Scale for Game-Based Learning Strategies, originally developed by Manzano-León et al. (2021) and adapted into Turkish by Küçükibiş and Eskiler (2022). The scale evaluates students' motivation across various dimensions related to game-based learning environments using Likert-type items. A higher total score indicates a higher level of motivation toward learning through gamification.

IPD SHARING:
Plan to Share IPD: No